CLINICAL TRIAL: NCT00949247
Title: Docetaxel, Carboplatin, Trastuzumab and Bevacizumab (TCH+B) For Early-Stage HER-2/Neu(+) Breast Cancer and Bone Marrow Micrometastases
Brief Title: Docetaxel,Carboplatin,Trastuzumab and Bevacizumab for Breast Cancer and Bone Marrow Micrometastases
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4108
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Trastuzumab; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel,Carboplatin,Trastuzumab and Bevacizumab (Experimental)
  Interventions: Biological: bevacizumab; Biological: trastuzumab; Drug: carboplatin; Drug: docetaxel; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, treatment modifications may apply according to response.
Biological: trastuzumab — Trastuzumab IV over 30-90 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, treatment modifications may apply according to response.
Drug: carboplatin — Carboplatin IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, treatment modifications may apply according to response.
Drug: docetaxel — Docetaxel IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, treatment modifications may apply according to response.
Other: laboratory biomarker analysis — Tumor tissue and bone marrow samples may be collected for further laboratory analysis.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy together with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This clinical trial is studying how well giving docetaxel and carboplatin together with trastuzumab and bevacizumab works in treating patients with stage I, stage II, or stage III breast cancer and bone marrow micrometastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response in patients with HER2/neu-positive stage I-III breast cancer and bone marrow micrometastases treated with docetaxel, carboplatin, trastuzumab, and bevacizumab.

Secondary

* Investigate the specific contribution of VEGF and CXCL-12 (SDF-1) signaling to bone marrow support of HER2/neu-positive breast cancer cells.
* Evaluate growth factor and chemokine expression profiles to investigate the potential correlation of expression with patient outcome and frequency of tumor cell clusters (mammospheres with tumor stem cell phenotype) in microenvironment supported cultures.

OUTLINE: Patients receive docetaxel IV, carboplatin IV, and bevacizumab IV over 30-90 minutes on day 1 and trastuzumab IV over 30-90 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, treatment modifications may apply according to response.

Tumor tissue and bone marrow samples may be collected for further laboratory analysis.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria

* Patient with biopsy-proven primary stage I-III infiltrating adenocarcinoma of the breast.
* HER-2/neu (+) as determined by either IHC (3+) or FISH (≥ 2.2-fold amplification).
* Age ≥ 18 years.
* ECOG performance status 0-1.
* Negative CT C/A/P and TBBS.
* LVEF > 50% by MUGA or echocardiogram performed within 28 days prior to enrollment
* Positive BM aspirate for BC micrometastases by CLIA-certified laboratory.
* Adequate hematologic, hepatic, and renal function. All tests must be obtained ≤ 4 weeks prior to randomization.

  * Hematologic: Absolute neutrophil count > 1,500/mm3 Hemoglobin > 10.0 g/dl Platelet count > 100,000/mm3.
  * Hepatic: Total bilirubin must be within normal limits. Transaminases (AST and/or ALT) may be < 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is < ULN, or alkaline phosphatase may be < 4 x ULN if transaminases are < ULN
  * Renal: Normal creatinine and BUN; if abnormal, calculated creatinine clearance must be> 60 mg/dL
* Patients must be disease-free of prior invasive malignancies for ≥ 5 years, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Surgery: all patients must have completed surgery with sentinel and/or axillary lymph node dissection according to participating institutional guidelines.
* Women of childbearing potential must have a negative pregnancy test and must be willing to consent to using an accepted and effective barrier form method of contraception while on treatment and for a reasonable period thereafter.
* Patients must provide written informed consent.
* Note: Hormonal therapy: patients with ER+ and/or PR+ tumors may receive concurrent hormonal therapy according to participating institutional guidelines. The choice of hormonal therapy is at the discretion of the treating physician.
* Note: Radiation therapy: patients receiving adjuvant radiation therapy to the involved breast (after partial mastectomy) or chest wall (after mastectomy) may receive concurrent trastuzumab and bevacizumab therapy.

Exclusion Criteria

* Known metastatic BC.
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Pregnant or lactating women.
* Prior chemotherapy, hormonal therapy, trastuzumab and bevacizumab therapy.
* History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
* Ejection fraction <50% or below the lower limit of the institutional normal range, whichever is lower.
* Hypersensitivity to trial medications.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest.
* Active or uncontrolled infection.
* Psychiatric, addictive, or any disorder that compromises the ability to give informed consent to participate in or to comply with the requirements of the study.

Bevacizumab-Specific Exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Known CNS disease
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either
* Urine protein:creatinine (UPC) ratio >/= 1.0 at screening OR
* Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential
* History of stroke or transient ischemic attack at any time
* History of myocardial infarction or unstable angina within 12 months of study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have a complete response in bone marrow. | at 4 weeks after completing 6 courses of therapy

SECONDARY OUTCOMES:
Specific contribution of VEGF and CXCL-12 (SDF-1) signaling to bone marrow support of HER2/neu-positive breast cancer cells | pre- and post-treatment
Potential correlation of growth factor and chemokine expression with patient outcome and frequency of tumor cell clusters (mammospheres with tumor stem cell phenotype) in microenvironment supported cultures | pre- and post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Baar, MD, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center; Thomas Budd, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Hospitals Monarch, Mayfield Heights, Ohio
  - University Hospitals Chagrin Highlands Medical Center, Orange, Ohio
  - University Hospitals Westlake, Westlake, Ohio